CLINICAL TRIAL: NCT06491108
Title: Vardenafil Versus Tadalafil Versus Tamsulosin in Patients With Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia: A Prospective Randomized Study.
Brief Title: Medications for Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hazem Bashir Ali Mohamed Baz, Urology resident at Tanta university hospitals, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vardenafil for BPH / LUTS
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Enlarged Prostate With Lower Urinary Tract Symptoms
MeSH Terms: interventions — Vardenafil Dihydrochloride; Tablets

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vardenafil in patients with lower urinary tract symptoms secondary to benign prostatic hyperplasia (Experimental): 50 patients will take Vardenafil 5 mg tabs twice daily and will be assessed at 4th week and 12th week. Treatment efficacy will be assessed by a change in pre and post treatment Q-max, PVR (post void residual urine), IPSS, (International Prostate Symptom Score) and Sexual Health Inventory for Men (SHIM) with monitoring any side effects
  Interventions: Drug: Vardenafil 5 Mg Oral Tablet
- Tadalafil in patients with lower urinary tract symptoms secondary to benign prostatic hyperplasia (Active Comparator): 50 patients will take Tadalafil 5 mg tabs once daily and will be assessed at 4th week and 12th week. Treatment efficacy will be assessed by a change in pre and post treatment Q-max, PVR (post void residual urine), IPSS, (International Prostate Symptom Score) and Sexual Health Inventory for Men (SHIM) with monitoring any side effects
  Interventions: Drug: Vardenafil 5 Mg Oral Tablet
- Tamsulosin in patients with lower urinary tract symptoms secondary to benign prostatic hyperplasia (Active Comparator): 50 patients will take Tamsulosin 0.4 mg tabs once daily and will be assessed at 4th week and 12th week. Treatment efficacy will be assessed by a change in pre and post treatment Q-max, PVR (post void residual urine), IPSS, (International Prostate Symptom Score) and Sexual Health Inventory for Men (SHIM) with monitoring any side effects
  Interventions: Drug: Vardenafil 5 Mg Oral Tablet

INTERVENTIONS:
Drug: Vardenafil 5 Mg Oral Tablet — Comparing safety and efficacy of Vardenafil 5 mg twice oral daily versus established drugs e.g.Tadalafil 5mg and Tamsulosin 0.4 mg once oral daily in terms of (voiding function, sexual function and quality of life) in the management of moderate BPH related LUTS (benign prostatic hyperplasia related lower urinary tract syptoms )
  Other Names: Vardenafil 5 mg

SUMMARY:
The main objective of this prospective randomized controlled study is to compare safety and efficacy of Vardenafil versus Tadalafil versus Tamsulosin in terms of (voiding function, sexual function and quality of life) in the management of moderate BPH related LUTS.

DETAILED DESCRIPTION:
This is prospective randomized controlled study that will be conducted on men with BPH related LUTS amenable to medical treatment at Urology Department, Faculty of Medicine, Tanta University - Egypt after having their written informed consent.

The study is planned to include 150 patients in the study period from April 2024 to April 2025. Each enrolled patient must complete 12 weeks on medication with strict scheduled follow up.

Inclusion criteria:

Sexually active patients with moderate BPH related LUTS amenable to medical treatment and completed 12 weeks follow up period.

Exclusion criteria:

Indication for combined therapy in patients who have moderate to severe LUTS and an increased risk of disease progression (e.g. prostate volume more than 40 ml) or patients in need for anti-muscarinic for predominant storage symptoms.

Indication for surgical intervention:

Medically complicated patients:

Cardiac patients, unstable angina, recent myocardial infarction (<3months), hypotension.

Concomitant uses (potassium channel openers, alpha 1 blockers, nitrates). Stroke since less than 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Sexually active patients .
2. ModerateBPH related LUTS ( bengin prostatic hyperplasia related lower urinary tract symtoms ) i.e: (international prostatic symptom score 8 to 19 : the higher score is the worse symptoms ).
3. Patients accepted medical treatment and completed 12 weeks on medical treatment and strict follow up .

Exclusion Criteria:

1. Indication for combined therapy as prostate size over 40 gm .
2. Gross hematuria.
3. Refractory urine retention .
4. Bilateral hydro-ureteronephrosis or renal insufficiency secondary to bengin prostatic hyperplasia.
5. Bladder diverticula or calculi .
6. History of bladder or prostate cancer.
7. Unwilling patients to medical therapy.
8. History of pelvic surgery or urethral stricture.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male gender
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
International prostate symptom score (IPSS total score) | 3 months
  Change in pre and post treatment condition (IPSS : international prostate symptom score - decresing in the score equals improving the symptoms )
The maximum urinary flow rate (Q-max) | 3 months
  Change in pre and post treatment condition (increasing at Q-max equals improving the symptoms )

SECONDARY OUTCOMES:
Sexual Health Inventory for Men (SHIM) | 3 months
  Change in pre and post treatment condition (SHIM: Sexual Health Inventory for Men - increasing in the score equals improving the symptoms )

CONTACTS AND LOCATIONS:
Overall Officials: Hazem B. Baz, M.B.B.Ch, Principal Investigator — Tanta University
Locations (1):
- Faculity of medicine - Tanta university, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagasubramanian S, John NT, Antonisamy B, Mukha RP, Jeyachandra Berry CS, Kumar S, Devasia A, Kekre NS. Tamsulosin and placebo vs tamsulosin and tadalafil in male lower urinary tract symptoms: a double-blinded, randomised controlled trial. BJU Int. 2020 May;125(5):718-724. doi: 10.1111/bju.15027. Epub 2020 Feb 27. PMID 32012409
- [Result] Stief CG, Porst H, Neuser D, Beneke M, Ulbrich E. A randomised, placebo-controlled study to assess the efficacy of twice-daily vardenafil in the treatment of lower urinary tract symptoms secondary to benign prostatic hyperplasia. Eur Urol. 2008 Jun;53(6):1236-44. doi: 10.1016/j.eururo.2008.01.075. Epub 2008 Feb 4. PMID 18281145